CLINICAL TRIAL: NCT05354531
Title: Outcome of the Anterior Subcutaneous Internal Fixator (INFIX) for Pelvic Ring Disruptions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Kyrillos Talaat saadallah abdelshahid, Professor Doctor Osama Farouk Head of trauma unit in department of orthopedic surgery Assiut university, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: INFIX
Record Dates: First submitted 2022-03-01; First posted 2022-04-29 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Pelvic Fracture
Keywords: pelvic ring fractures; INFIX
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Intervention Model Description: One group of 20 cases should be managed by INFIX for their pelvic ring disruption
Masking Description: Those previously mentioned cases should be assessed clinically and radiologically
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- INFIX group (Experimental): Those group of cases will be managed by INFIX for their pelvic ring disruption
  Interventions: Procedure: anterior subcutaneous internal fixator ( INFIX)

INTERVENTIONS:
Procedure: anterior subcutaneous internal fixator ( INFIX) — INFIX was invented based upon the same biomechanical principle as the traditional external fixator, but it is placed subcutaneously. It proved to be stiffer than the traditional external fixator, and at the same time eliminates the open pin tracts, which increased the infection rate and nursing care

SUMMARY:
With a prospective case series study of 15 patients The aim of this study is to estimate the clinical outcomes in patients with unstable anterior pelvic ring fractures ( B&C ) after treatment with (INFIX)

DETAILED DESCRIPTION:
Unstable pelvic ring fractures are usually associated with high energy trauma. They account for about 1.5-3.9% of all fractures, but they have a high rate of morbidity and mortality. Although the posterior pelvic ring provides the main stability (60%), the anterior ring still account for 40% of stability fracture pelvis B &C according to tiles classification require fixation of the anterior ring or anterior-posterior ring simultaneously.

The external fixator is the most widely used treatment for initial and temporary stabilization of anterior pelvic ring injury, especially in emergency situations. It can be quickly placed and can easily stabilize the disrupted pelvic ring and decrease pelvic cavity haemorrhage. However, many clinical complications associated with the external fixator have been reported, including wound infection, loosening of the fixator, and impingement on the skin.

Moreover, the anterior pelvic external fixator limits patients' daily activities, such as sitting, lying in the lateral position, rolling over, and sexual intercourse

Recently, anterior subcutaneous internal fixator (INFIX) was proposed by several scholars to treat anterior pelvic ring injury.

INFIX was invented based upon the same biomechanical principle as the traditional external fixator, but it is placed subcutaneously. It proved to be stiffer than the traditional external fixator, and at the same time eliminates the open pin tracts, which increased the infection rate and nursing care .

INFIX was initially designed as an alternative to the external fixator, but recently its indications have been expanded and multiple complications have been reported.

ELIGIBILITY:
Inclusion Criteria:

* skeletally mature patient.
* type B2 / B3 & C1 pelvic fracture.
* open book B1 fracture with urogenital disruption.
* Patient with fatty tissue that cover pubic bones enable insertion of the rod.
* if there is a contraindication to Anterior symphyseal plating.

Exclusion Criteria:

* associated comorbidities preventing surgery.
* pelvic fracture associated with iliac bones fracture
* combined pelvis and acetabulum fracture.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-03-02 (Actual); Primary Completion 2025-03-11 (Actual); Study Completion 2025-03-11 (Actual)

PRIMARY OUTCOMES:
Majeed score | After 3 months
  Majeed rating scale will be used to evaluate the functional outcome. Patients will be followed up by phone or at the clinic. functional recovery will be scored by asking the rating scale questions. These questions including the subjective feelings of pain, return to the work, the feelings of sitting, sexual intercourse, standing, walking distance, and the condition of gait. The aggregate score will be classified as excellent (>85), good (70-84), fair (55-69), or poor (<55).

SECONDARY OUTCOMES:
Time to surgery | Within the first week
  We will assess the time taken for the patient to be in the operation
Radiology dose | Within the first week
  Sum of radiology dose taken intraoperatively
Procedure time | Within the first week
  Time taken intraoperatively
Incidence and rate of adverse events | After 6 months
  Any complications or problems should be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Osama Farouk, Prof, Study Chair — Orthopedic surgery department ,Assiut university
Locations (2):
- Egypt (2):
  - Orthopedic and trauma department Assiut university, Asyut
  - Orthopedic and traumatology department Assiut university hospital, Asyut

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Merriman DJ, Ricci WM, McAndrew CM, Gardner MJ. Is application of an internal anterior pelvic fixator anatomically feasible? Clin Orthop Relat Res. 2012 Aug;470(8):2111-5. doi: 10.1007/s11999-012-2287-6. PMID 22383020